CLINICAL TRIAL: NCT02172365
Title: Retrospective Analysis of Treatment Outcomes of Allogeneic Stem Cell Transplantation for Chronic Myeloid Leukemia After TKI Failure
Brief Title: Allogeneic SCT for CML, TKI Failure After TKI Failure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN 14-7493-AE
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; Allogeneic hematopoietic cell transplantation; Tyrosine kinase inhibitor; TKI failure
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will evaluate the outcomes of allogeneic stem cell transplantation which is the only curative treatment modality in the patients with chronic myeloid leukemia after failing tyrosine kinase inhibitor therapy. However, any update was not reported on the transplant outcomes in the patients failed TKI therapy, thus necessitating update of this data. Also, the European Group for Blood and Marrow Transplantation (EBMT) risk score is still of value, but insufficient numbers of patients have been transplanted in recent years and after TKI therapy to allow a robust reanalysis. Our study hypothesis is that allogeneic SCT treatment modality can rescue CML patients who failed TKI therapy due to resistance or to intolerance with improved survival and long-term outcomes. Also, another hypothesis will be examined if the EBMT risk score proposed pre-imatinib era can reproduce similar prognostic risk stratification of long-term outcomes in the patients treated with TKI.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation (SCT) remains the only currently available treatment that can render patients durably molecularly negative, but the associated procedural-related morbidity and mortality remain a major deterrent.

Currently the followings are accepted as reasonable indication for allogeneic SCT for CML: failure to 2nd generation tyrosine kinase inhibitor (2GTKI) after imatinib failure, 2GTKI frontline failure, or any patients meeting the criteria of failure such as development of additional cytogenetic abnormality (ACA), clonal evolution in ph neg clone, development of mutation and loss of CCyR as well as any advanced disease stage including accelerated or blastic phase. However, insufficient numbers of patients have been transplanted in recent years and after TKI therapy, thus necessitating update of this data.

The EBMT risk score has been used for a decade for the decision making of transplantation in the pre-imatinib era. However, it has never been re-evaluated in a larger cohort of CML patients treated with TKIs prior to SCT then received alloSCT, thus requiring to be reanalysed for its prognostic implication on long-term survival.

As mentioned above, any update was not reported on the transplant outcomes in the patients failed TKI therapy, thus necessitating update of this data. Also, the EBMT risk score2 is still of value, but insufficient numbers of patients have been transplanted in recent years and after TKI therapy to allow a robust reanalysis.

This is retrospective study. The medical records will be reviewed retrospectively. The treatment outcomes such as complete cytogenetic response (CCyR), major molecular response (MMR), molecular response at 4.5 log reduction (MR4.5), treatment failure (TF), progression free survival (PFS) and overall survival (OS) will be estimated using Kaplan-Meier method. The CCR will be defined as 0% of Ph+ metaphase cells in the marrow or less than 1% by international scale using BCR-ABL1 transcript polymerase chain reaction (PCR) test. The MMR is defined as lower than or equal to a 0.1%IS of BCR-ABL1 fusion gene transcripts, and MR4.5 is defined as 0.0032%IS BCR-ABL1 transcript level, equivalent to a 4.5 log reduction of BCR-ABL1 transcript level. Time to treatment failure (TTF) is defined as the interval between allogeneic SCT and the occurrence of events that indicated that CML has relapsed including primary hematologic resistance, cytogenetic resistance, loss of CCyR, development of ABL tyrosine kinase domain mutation, clonal evolution and progression to accelerated phase (AP) or blastic crisis (BC). Death is considered as censored for TTF. Time to PFS is defined as the interval between transplantation and confirmation of progression to AP or BC or death from any cause, while OS was calculated from transplantation until the date of death from any cause or of latest follow-up.

Pre-transplant characteristics and transplant procedure data will be also collected including the age, disease stage, diagnosis/transplant date, donor type and gender match. Summary of treatment outcomes following previous TKI therapies will be also collected. Post-transplant events such as graft-versus-host disease (GVHD) and progression of CML will be also collected.

No study intervention.

Assessment of Efficacy:

Cytogenetic responses were categorized as complete (0% Ph+ cells in marrow by conventional cytogenetics), partial (1% to 34% Ph+ cells in marrow), or minor (35% to 90% Ph+ cells in marrow). A major cytogenetic response (MCyR) was defined as the sum of CCyR and partial cytogenetic response (i.e. 0% - 35% Ph+ cells in marrow). Major molecular response (MMR) was defined as lower than or equal to a 0.1%IS of BCR-ABL1 fusion gene transcripts, and molecular response 4.5 (MR4.5) was defined as 0.0032%IS BCR-ABL1 transcript level, equivalent to a 4.5 log reduction of BCR-ABL1 transcript level.

Time to treatment failure (TTF) is defined as the interval between allogeneic SCT and the occurrence of events that indicated that CML has relapsed including primary hematologic resistance, cytogenetic resistance, loss of CCyR, development of ABL tyrosine kinase domain mutation, clonal evolution and progression to accelerated phase (AP) or blastic crisis (BC). Death is considered as censored for TTF. Time to PFS is defined as the interval between transplantation and confirmation of progression to AP or BC or death from any cause, while OS was calculated from transplantation until the date of death from any cause or of latest follow-up.

Statistical analysis:

The list of CML patients will be utilized for this retrospective study. Study ID, gender, disease characteristics at the time of diagnosis, details of treatment, detailed response to treatment, resistance or intolerance and long-term outcomes will be retrospectively reviewed.

Study endpoints will be analyzed with respect to complete cytogenetic response (CCR), major/complete molecular response (MMR/CMR), loss of response, resistance, progression to advance disease and death. The cumulative incidence of CCR, MMR and CMR will be estimated and compared using the approach proposed by Gray (Gray, 1988). Overall survival will be analyzed using the Kaplan-Meier method and compared using the log-rank test. Loss of response, resistance and failure-free survival will be analyzed using the test for cumulative incidence to account for competing risk events. Baseline characteristics, including Sokal score, age, gender, disease stage, will be adopted as surrogates for further response, progression free and overall survival following transplantation. For the EBMT risk score, age of the patient, stage of the disease at transplant, time from diagnosis (<12 months vs > 12months), donor type, and donor recipient gender combination will be used for the calculation. The transplant outcomes will be compared according to the EBMT risk score.

P-values of less than 0.05 will be considered statistically significant. Hazard ratios (HR) and 95% confidence intervals (CI) will be estimated with a predetermined reference risk of 1.0. The EZR software will be used for the statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with allogeneic stem cell transplantation (SCT) since 2000 till 2013 for any of tyrosine kinase inhibitor (TKI) failure due to resistance or intolerance during chronic myeloid leukemia (CML) management with tyrosine kinase inhibitor

Exclusion Criteria:

* Any CML patients not previously treated with TKI therapy prior to allogeneic stem cell treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with allogeneic stem cell transplantation (SCT) since 2000 till 2013 for any of tyrosine kinase inhibitor (TKI) failure due to resistance or intolerance during chronic myeloid leukemia (CML) management with tyrosine kinase inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2014-03-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival following allogeneic SCT for CML after TKI failure. | at 3 years
  Overall survival will be calculated from transplantation until the date of death from any cause or of latest follow-up

SECONDARY OUTCOMES:
Failure free survival following allogeneic SCT for CML after TKI failure | at 3 years
  Time to failure free survival is defined as the interval between transplantation and treatment failure. Treatment failure will be defined as primary hematologic resistance, cytogenetic resistance, loss of CCyR, development of ABL tyrosine kinase domain mutation, clonal evolution and progression to accelerated phase (AP) or blastic crisis (BC).
Relapse following allogeneic SCT for CML after TKI failure | at 3 years
  Relapse will be defined as confirmation of progression to AP or BC.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Baccarani M, Deininger MW, Rosti G, Hochhaus A, Soverini S, Apperley JF, Cervantes F, Clark RE, Cortes JE, Guilhot F, Hjorth-Hansen H, Hughes TP, Kantarjian HM, Kim DW, Larson RA, Lipton JH, Mahon FX, Martinelli G, Mayer J, Muller MC, Niederwieser D, Pane F, Radich JP, Rousselot P, Saglio G, Saussele S, Schiffer C, Silver R, Simonsson B, Steegmann JL, Goldman JM, Hehlmann R. European LeukemiaNet recommendations for the management of chronic myeloid leukemia: 2013. Blood. 2013 Aug 8;122(6):872-84. doi: 10.1182/blood-2013-05-501569. Epub 2013 Jun 26. PMID 23803709
- [Background] Gratwohl A, Hermans J, Goldman JM, Arcese W, Carreras E, Devergie A, Frassoni F, Gahrton G, Kolb HJ, Niederwieser D, Ruutu T, Vernant JP, de Witte T, Apperley J. Risk assessment for patients with chronic myeloid leukaemia before allogeneic blood or marrow transplantation. Chronic Leukemia Working Party of the European Group for Blood and Marrow Transplantation. Lancet. 1998 Oct 3;352(9134):1087-92. doi: 10.1016/s0140-6736(98)03030-x. PMID 9798583
- [Background] Jabbour E, Cortes J, Santos FP, Jones D, O'Brien S, Rondon G, Popat U, Giralt S, Kebriaei P, Jones RB, Kantarjian H, Champlin R, de Lima M. Results of allogeneic hematopoietic stem cell transplantation for chronic myelogenous leukemia patients who failed tyrosine kinase inhibitors after developing BCR-ABL1 kinase domain mutations. Blood. 2011 Mar 31;117(13):3641-7. doi: 10.1182/blood-2010-08-302679. Epub 2010 Dec 14. PMID 21156844
- [Background] Nicolini FE, Basak GW, Soverini S, Martinelli G, Mauro MJ, Muller MC, Hochhaus A, Chuah C, Dufva IH, Rege-Cambrin G, Saglio G, Michallet M, Labussiere H, Morisset S, Hayette S, Etienne G, Olavarria E, Zhou W, Peter S, Apperley JF, Cortes J. Allogeneic stem cell transplantation for patients harboring T315I BCR-ABL mutated leukemias. Blood. 2011 Nov 17;118(20):5697-700. doi: 10.1182/blood-2011-07-367326. Epub 2011 Sep 16. PMID 21926354
- [Background] Saussele S, Lauseker M, Gratwohl A, Beelen DW, Bunjes D, Schwerdtfeger R, Kolb HJ, Ho AD, Falge C, Holler E, Schlimok G, Zander AR, Arnold R, Kanz L, Dengler R, Haferlach C, Schlegelberger B, Pfirrmann M, Muller MC, Schnittger S, Leitner A, Pletsch N, Hochhaus A, Hasford J, Hehlmann R; German CML Study Group. Allogeneic hematopoietic stem cell transplantation (allo SCT) for chronic myeloid leukemia in the imatinib era: evaluation of its impact within a subgroup of the randomized German CML Study IV. Blood. 2010 Mar 11;115(10):1880-5. doi: 10.1182/blood-2009-08-237115. Epub 2009 Nov 18. PMID 19965667